CLINICAL TRIAL: NCT02008786
Title: The Effects of Statin and Angiotensin-converting Enzyme Inhibitor on Coronary Flow Reserve, indEx of Microcirculatory Resistance, and Symptoms in Patients With Spontaneous Coronary Artery Dissection (SAFER-SCAD) Study
Brief Title: Statin and Angiotensin-converting Enzyme Inhibitor on Symptoms in Patients With SCAD
Acronym: SAFER-SCAD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Cardiology Research UBC (Other)
Responsible Party: Principal Investigator, Dr. Tara Sedlak, Cardiologist, Cardiology Research UBC
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAFER-SCAD
Record Dates: First submitted 2013-12-07; First posted 2013-12-11 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Dissection, Spontaneous
Keywords: Coronary Artery Dissection, Spontaneous; Angina
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous; Angina Pectoris | interventions — Ramipril; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin, placebo (Experimental): rosuvastatin 10-20mg daily or placebo (suggested dose of 10mg for Asians, and 20mg for others)
  Interventions: Drug: rosuvastatin; Drug: placebo
- Ramipril, placebo (Experimental): ramipril (starting dose of ramipril at 5mg daily titrating up to 10mg daily at 1 week if tolerated) versus placebo
  Interventions: Drug: ramipril; Drug: placebo

INTERVENTIONS:
Drug: ramipril — 5-10mg (starting dose 5mg titrating up to 10mg if tolerated after 1 week)
  Other Names: Altace
  Arms: Ramipril, placebo
Drug: rosuvastatin — 10-20mg (suggested dose 10mg for Asians, 20mg for everyone else)
  Other Names: crestor
  Arms: Rosuvastatin, placebo
Drug: placebo — Placebo

SUMMARY:
An emerging cause of heart attack in young women is a dissection (or tear) in the coronary arteries. Many of these young women continue to have chest pain long after the tear has healed and this is thought to be due to problems with their small blood vessels of the heart (or microcirculation). We want to determine whether commonly used medications for coronary artery disease including statins (for cholesterol) and angiotensin-converting enzyme inhibitors (for blood pressure) reduce chest pain and improve small vessel function in these patients.

DETAILED DESCRIPTION:
In patients with spontaneous coronary artery dissection (SCAD), many continue to have ongoing signs and symptoms of ischemia after the dissection has healed. Further, 1 in 5 women will experience recurrent SCAD in long-term follow-up. To date, no study has investigated the pathophysiologic mechanism behind ongoing symptoms or recurrence of SCAD, but microvascular coronary dysfunction (MCD) has been suggested. Coronary reactivity testing (CRT) is an invasive procedure currently being done in MCD patients as the gold standard technique. In particular, a coronary flow reserve (CFR) < 2.5 has been shown to be both diagnostic of the condition and prognostic of a 2 fold increased risk of cardiac events. Please see below for a detailed description of CRT. In brief, a dual temperature and pressure sensor tipped wire by Radi Medical Systems (St Jude Medical, St Paul, MN) will be placed into the dissected and non-dissected coronary arteries of the patient. This will measure CFR by thermodilution and will also allow the measurement of the index of microcirculatory resistance (IMR). IMR has been found to correlate well with true microvascular resistance.

In addition to a lack of diagnostic strategies, there is a paucity of research into therapeutic strategies. Most women are conservatively managed with medications, however, there is no consensus as to which pharmacologic therapies should be used. Case reports have suggested benefit with antiplatelet agents (e.g. aspirin) and beta-blockers (reduction of arterial wall shear stress). To date no study has investigated the effects of statins or Angiotensin Converting Enzyme Inhibitors (ACEIs) in SCAD patients. Both agents have been studied in the MCD population and been found to reduce angina frequency and improve CFR after 16 weeks.

Purpose:

To measuring the CFR and IMR in 40 SCAD patients with ongoing chest pain who are at least 3 months from their dissection to determine the proportion with microvascular dysfunction and to investigate prospectively whether the addition of an ACEI or a statin to usual care in patients with ongoing chest pain and a CFR <3.0 improves chest pain frequency by Seattle Angina Questionnaire (SAQ) at 16 weeks compared to placebo.

Hypothesis:

We hypothesize that the average CFR in patients at least 3 months out from their SCAD will be <2.5 and that their IMR will be abnormal. Further, we hypothesize that the addition of either an ACEI and/or statin will improve chest pain frequency by at least 20 points on the SAQ at 16 weeks compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Any woman with prior SCAD who is at least 3 months out from her SCAD and has ongoing symptoms of chest pain.
* Females of child-bearing age must have a negative pregnancy test at enrollment
* Coronary Flow Reserve(CFR) < 3.0

Exclusion Criteria:

* Renal dysfunction with Glomerular Filtration Rate <50 ml/min
* Patients not willing to undergo coronary angiography
* Patients with a prior intolerance or allergy to rosuvastatin or ramipril
* Inability to perform CRT or CFR >3.0
* Obstructive coronary artery disease (stenosis >50% in any artery) or residual dissection >50% with distal flow abnormalities

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06; Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Angina frequency domain of the SAQ | 16 weeks after each intervention
  Angina frequency domain of the SAQ, collected at baseline and after each intervention to assess angina frequency change over time. We hypothesize that mean SAQ will improve by at least 20 points in each treatment group compared to placebo.

SECONDARY OUTCOMES:
Acute coronary syndrome or hospitalization for angina | 1 year
  As a secondary objective, to evaluate whether ACEI or statin versus placebo reduces the combined endpoint of acute coronary syndrome (ACS) or hospitalization for angina at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tara Sedlak, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada